CLINICAL TRIAL: NCT02672163
Title: Epicardial Delivery of Autologous Atrial Appendage Micrografts During Coronary Artery Bypass Surgery - Safety and Feasibility Study
Brief Title: Autologous Atrial Appendage Derived Cells in the Treatment of Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Ari Harjula, Professor, Clinical research, Helsinki University Central Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 180/13/03/02/2013
Record Dates: First submitted 2015-12-28; First posted 2016-02-03 (Estimated); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Heart Failure
Keywords: autologous micrografts; heart failure; coronary artery bypass surgery; cell therapy; atrial appendage; epicardial cell delivery
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AACD-Therapy group (Experimental): 6 patients are recruited to the AADC-therapy group. Autologous atrial appendage derived cells (AADCs) are harvested from the appendage tissue removed during the venal cannulation of bypass. The cells and their extracellular matrix are placed with tissue clue to Cormatrix-sheet and further on top of the myocardium in the area of infarction scar. The procedure is done simultaneously with CABG surgery. The patients will be carefully monitored after the operations and cardiac MRI and echocardiogram will be performed previously to surgery as well as during the follow ups.
  Interventions: Procedure: CABG surgery; Procedure: AADC therapy
- Control group (Active Comparator): 20 patients are recruited to form the control group. They are patients scheduled for elective CABG surgery and they meet the same inclusion and exclusion criteria as the therapy group. There patients are followed as the hospital protocol with out any additional imagination or blood tests.
  Interventions: Procedure: CABG surgery

INTERVENTIONS:
Procedure: CABG surgery — Elective CABG surgery
Procedure: AADC therapy — Atrial appendage derived cells are placed on the site of a infarct scar with matrix sheet
  Arms: AACD-Therapy group

SUMMARY:
This study aims to evaluate the safety and clinical feasibility of epicardially delivered autologous atrial appendage micrografts in the treatment of heart failure. The micrografts consisting atrial-derived cells and their extracellular matrix, are placed on an infarction scar during CABG surgery.

DETAILED DESCRIPTION:
The atrial appendages are a tissue reservoir for cardiomyocyte stem and precursor cells. During coronary artery bypass graft (CABG) surgery part of the right atrial appendage can be excised upon insertion of the right atrial cannula of the heart-lung machine. This study aims to address the surgical feasibility and patient safety of epicardially delivered atrial appendage micrografts during CABG surgery.

Autologous cardiac cells are harvested from right atrial appendage during CABG of six patients. Micrografts consisting atrial appendage-derived cells (AADCs) and their extracellular matrix (ECM) of the atrial appendage are mechanically processed. The cells are placed on a tissue-engineered sheet with fibrin gel and tissue clue and further delivered epicardially on top of a infarction scar. Parameters including echocardiography reflecting cardiac insufficiency are studied pre- and post-operatively as well as at three and six months of the follow-up. Cardiac functional magnetic resonance imaging is performed preoperatively and at six-months follow-up. 20 patients will be recruited to serve as a control group. They are scheduled for elective CABG and are treated according to the normal hospital protocol, without the ECM sheet.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained
* Left ventricular ejection fraction (LVEF) between ≤50% and ≥15%
* New York Heart Association (NYHA) Class II-IV heart failure symptoms

Exclusion Criteria:

* Heart failure due to left ventricular outflow tract obstruction
* History of life-threatening and possibly repeating ventricular arrhythmias or resuscitation, or an implantable cardioverter-defibrillator
* Stroke or other disabling condition within 3 months before screening
* Severe valve disease or scheduled valve surgery
* Renal dysfunction (GFR <84 ml/min/1.73m)
* Other disease limiting life expectancy
* Contraindications for coronary angiogram or MRI
* Participation in some other clinical trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-02; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Safety; need for vasoactive medication | 6 months
  For assessing haemodynamics during the operation and at the intensive care unit
Safety; cardiac index in l/min/m | 6 months
  For assessing haemodynamics during the operation and at the intensive care unit
Safety; hemoglobin in g/l | 6 months
  For assessing haemodynamics during the operation and at the intensive care unit
Safety; oxygen saturation in the pulmonary arterial blood (SvO2) in % | 6 months
  For assessing haemodynamics during the operation and at the intensive care unit
Safety; serum potassium level in mmol/l | 6 months
  For assessing haemodynamics during the operation and at the intensive care unit
Safety; blood glucose level in mmol/l | 6 months
  For assessing haemodynamics during the operation and at the intensive care unit
Safety; Left ventricular ejection fraction (EF) in % | 6 months
  For assessing cardiac function during and after the operation by echocardiogram
Safety; pericardial effusion in mm | 6 months
  For assessing cardiac function after the operation by echocardiogram
Safety: telemetric monitoring of rhythm | 6 months
  For assessing cardiac function after the operation
Feasibility: Success in completing the delivery of the cell sheet to the myocardium | 6 months
  Measured in 0= success, 1= no success
Feasibility: Waiting time in minutes for the cell sheet | 6 months
  Waiting time in minutes for the finished cell sheet to be placed on the myocardium after doing all the required anastomoses
Feasibility: Waiting time in minutes for the heart | 6 months
  Waiting time in minutes for the the heart after doing all the anastomoses and before the cell sheet is finished
Feasibility: Closing the right atrial appendage | 6 months
  Closing the right atrial appendage after removing the standardized tissue piece for preparing the cell sheet. According to the hospital protocol, appendage is closed with purse string suture. 0 = no additional suturing needed, 1 = additional suturing needed.

SECONDARY OUTCOMES:
Left ventricular wall thickness | 6 months
  Measured by MRI
Change in the amount of myocardial scar tissue | 6 months
  Measured by MRI
Change in left ventricular ejection fraction | 6 months
  Measured by MRI
Plasma concentrations of N-terminal pro-B-type natriuretic peptide (NT-proBNP) levels | 6 months
New York Heart Association class | 6 months
Days in hospital | 1 month
Changes in the quality of life. | 6 months
  measured by questionnaire
Change in movement and diastolic function of left ventricular wall | 6 months
  Measured by MRI
Local changes in systolic and diastolic function | 3 months
  Measured by echocardiogram

CONTACTS AND LOCATIONS:
Overall Officials: Ari Harjula, Prof, Study Director — Heart and Lung Center, Helsinki University Hospital
Locations (1):
- Annu Nummi, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lehtinen M, Patila T, Vento A, Kankuri E, Suojaranta-Ylinen R, Poyhia R, Harjula A; Helsinki BMMC Collaboration. Prospective, randomized, double-blinded trial of bone marrow cell transplantation combined with coronary surgery - perioperative safety study. Interact Cardiovasc Thorac Surg. 2014 Dec;19(6):990-6. doi: 10.1093/icvts/ivu265. Epub 2014 Aug 20. PMID 25142068
- [Background] Lehtinen M, Schildt J, Ahonen A, Nikkinen P, Lauerma K, Sinisalo J, Kankuri E, Vento A, Patila T, Harjula A; Helsinki BMMC Collaboration. Combining FDG-PET and 99mTc-SPECT to predict functional outcome after coronary artery bypass surgery. Eur Heart J Cardiovasc Imaging. 2015 Sep;16(9):1023-30. doi: 10.1093/ehjci/jev032. Epub 2015 Mar 9. PMID 25762563
- [Background] Lehtinen M, Patila T, Kankuri E, Lauerma K, Sinisalo J, Laine M, Kupari M, Vento A, Harjula A; Helsinki BMMC Collaboration. Intramyocardial bone marrow mononuclear cell transplantation in ischemic heart failure: Long-term follow-up. J Heart Lung Transplant. 2015 Jul;34(7):899-905. doi: 10.1016/j.healun.2015.01.989. Epub 2015 Feb 7. PMID 25797522
- [Background] Lampinen M, Vento A, Laurikka J, Nystedt J, Mervaala E, Harjula A, Kankuri E. Rational Autologous Cell Sources For Therapy of Heart Failure - Vehicles and Targets For Gene and RNA Therapies. Curr Gene Ther. 2016;16(1):21-33. doi: 10.2174/1566523216666160104141809. PMID 26725880
- [Derived] Nummi A, Mulari S, Stewart JA, Kivisto S, Teittinen K, Nieminen T, Lampinen M, Patila T, Sintonen H, Juvonen T, Kupari M, Suojaranta R, Kankuri E, Harjula A, Vento A; AADC consortium. Epicardial Transplantation of Autologous Cardiac Micrografts During Coronary Artery Bypass Surgery. Front Cardiovasc Med. 2021 Sep 14;8:726889. doi: 10.3389/fcvm.2021.726889. eCollection 2021. PMID 34595223
- [Derived] Nummi A, Nieminen T, Patila T, Lampinen M, Lehtinen ML, Kivisto S, Holmstrom M, Wilkman E, Teittinen K, Laine M, Sinisalo J, Kupari M, Kankuri E, Juvonen T, Vento A, Suojaranta R, Harjula A; AADC consortium. Epicardial delivery of autologous atrial appendage micrografts during coronary artery bypass surgery-safety and feasibility study. Pilot Feasibility Stud. 2017 Dec 20;3:74. doi: 10.1186/s40814-017-0217-9. eCollection 2017. PMID 29276625